CLINICAL TRIAL: NCT05490381
Title: Super-Selective Intra-Arterial Embolization of Hypervascular Head and Neck Tumors
Brief Title: Preoperative Embolization of Hypervascular Head and Neck Tumors to Improve Surgical Outcomes
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to no accruals and change in the standard of care for this population
Sponsor: University of Washington (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1121599; NCI-2022-05693 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00009998 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-10

CONDITIONS: Malignant Neoplasm in the Head and Neck; Metastatic Malignant Neoplasm in the Head and Neck
MeSH Terms: interventions — iodixanol; Polyvinyl Alcohol; Ethiodized Oil; Iodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (PVA, EOV, tumor vessel embolization) (Experimental): Patients receive iodixanol via injection and undergo diagnostic cerebral angiogram over 30 minutes. If the tumor blood supply is suitable, patients undergo tumor vessel embolization with PVA suspended in EOV and delivered via a catheter. Patients also undergo head and neck CT scans immediately after completion of tumor vessel embolization, and again between 2-3 months later.
  Interventions: Other: Iodixanol; Procedure: Angiogram; Procedure: Arterial Embolization; Drug: Polyvinyl Alcohol; Drug: Ethiodized Oil; Procedure: Computed Tomography; Other: Chart Abstraction

INTERVENTIONS:
Other: Iodixanol — Given via injection
  Other Names: Indixanol; OptiPrep; Visipaque
Procedure: Angiogram — Undergo diagnostic cerebral angiogram
Procedure: Arterial Embolization — Undergo tumor vessel embolization
  Other Names: TAE; Transarterial Embolization
Drug: Polyvinyl Alcohol — Given via catheter
  Other Names: 9002-89-5; Polydesis; Polyviol; Poval 420; PVA; Vinarol DT
Drug: Ethiodized Oil — Given via catheter
  Other Names: 8008-53-5; Ethiodol; iodized oil; Lipiodol
Procedure: Computed Tomography — Undergo head and neck CT scans
  Other Names: CAT Scan; Computed Axial Tomography; CT SCAN
Other: Chart Abstraction — Ancillary studies

SUMMARY:
This phase I trial tests whether embolization done prior to surgery (preoperative) will improve surgical outcomes in head and neck tumors with large amounts of blood vessels (hypervascular). Embolization is a minimally invasive surgical technique performed under angiographic (imaging of blood vessels) guidance. Embolization therapy injects tiny particles into the arteries feeding tumors to cut off their blood supply which may help improve outcomes by preventing blood loss during surgery, reducing surgical times, and shrinking tumors or reducing recurrence.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive iodixanol via injection and undergo diagnostic cerebral angiogram over 30 minutes. If the tumor blood supply is suitable, patients undergo tumor vessel embolization with polyvinyl alcohol (PVA) suspended in ethiodized oil (EOV) and delivered via a catheter. Patients also undergo head and neck computed tomography (CT) scans immediately after completion of tumor vessel embolization, and again between 2-3 months later.

After completion of study, patients are followed for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Primary or metastatic extra-axial tumor involving one or more anatomic structures in the head and neck
* Vascular supply from one or more branches of the external carotid artery
* Planned surgical resection
* All stages
* Extra-axial head and neck tumor greater than 1 cm in any dimension
* Confirmed by contrast-enhanced magnetic resonance imaging (MRI) or computed tomography (CT) of the head and/or neck
* Subjects who have undergone prior therapies are eligible
* Adults aged 18-80; no data outside this age range
* Minimum of 3-month life expectancy
* Estimated glomerular filtration rate (eGFR) greater than 30 mL/min/1.73 m^2
* Subjects must be non-pregnant at the time of angiographic intervention
* Resectable tumor as determined by the Tumor Board
* Medically stable at the time of the planned intervention, despite potential comorbidities
* In English or Spanish. All study materials have been professionally translated into Spanish

Exclusion Criteria:

* Recent hemorrhage or trauma
* Pregnancy
* Nursing mothers
* Contrast medium allergy
* Hypersensitivity or known allergy to ethiodized oil, poppy seeds, or poppy seed oil
* Uncontrolled or concurrent illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy is a contraindication to angiography outside of the emergency setting
* Active thyroid disease may be affected by iodinated products
* Subject is participating in another clinical trial at the enrollment of the study or duration of the study that can affect the treatment and outcome of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-21 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | Intraoperatively
  Defined as the volume of blood lost (mL) from skin incision to skin closure.

SECONDARY OUTCOMES:
Perioperative blood transfusion volume | Intraoperatively and until 48 hours postoperatively
  Defined as the volume (mL) of packed red blood cells infused.
Surgical procedure time | Time (minutes) from skin incision to skin closure
  Defined as the amount of time (minutes) from skin incision to skin closure.
Success of embolization | Directly after the embolization
  Defined as percent reduction in vascular blush from tumor supply vessels on catheter angiogram.
Adverse events (AE) related to angiography or embolization | Directly after embolization and for 24 hours post-embolization
  Defined as neurological deficit(s) on clinical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Walker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium; Do Lim, Study Director — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No